CLINICAL TRIAL: NCT06685146
Title: Investigating the Effect of Glucagon on Cognitive Function and Cerebral Glucose Metabolism in Humans: A Pilot Study
Brief Title: The Glucose-Independent Effects of Exogenous Glucagon on Insulin Secretion and Cognitive Function in Healthy Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolai Jacob Wewer Albrechtsen (Other)
Responsible Party: Sponsor-Investigator, Nicolai Jacob Wewer Albrechtsen, Principal Investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GluCoMet_pilotB
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Glucose Metabolism; Insulin Secretion
Keywords: Glucagon; Glucose Metabolism; Cognition; Glucose clamp; Insulin secretion; C-peptide
MeSH Terms: interventions — Glucose Clamp Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glucagon infusion followed by glucose-clamp (Experimental): The first study day is a 240 minutes infusion of glucagon (10ng/kg/min). The second study day is a 240 minutes infusion of glucose (20% w/v). The infusion rate of glucose will be adjusted continuously to match the levels of glucose measured on the glucagon study day.
  Interventions: Other: Glucagon Infusion; Other: Glucose clamp

INTERVENTIONS:
Other: Glucagon Infusion — A 240 minutes infusion of glucagon (10 ng/kg/min)
Other: Glucose clamp — A 240 minutes infusion of 20 % w/v glucose. The infusion rate of glucose will be adjusted continuously to match the levels of glucose measured on the glucagon study day.

SUMMARY:
In this study the investigators will investigate the glucose-independent effects of exogenous glucagon on insulin secretion and cognitive function in healthy subjects.

Subjects will participate in two study days. The first study day is with a 240-minute infusion of glucagon and the second study day is with an infusion of glucose (clamped to match the glucose levels measured during the glucagon infusion). During the study day, blood samples will be drawn frequently and cognitive testing will be performed.

The investigators will investigate glucagon's glucose-independent effects on insulin secretion and cognitive function by comparing plasma measures of C-peptide and cognitive test scores between the glucagon study day and the glucose clamp study day.

DETAILED DESCRIPTION:
Five-ten subjects with normal health will be included, and each subject will participate in two study days.

Participants will arrive after an overnight fast and will be placed in a hospital bed in a semi-recumbent position. In each antecubital vein an intravenous catheter will be placed; one for administration of glucagon or glucose and one for blood sampling. The first study day will be the glucagon study day. The blood measurements of glucose from the glucagon study day will be used for clamping the glucose levels during the glucose clamp study day.

Baseline blood samples will be drawn. At time 0 minutes the infusion of glucagon or glucose will be initiated. Glucagon will be infused at a rate of 10ng/kg/min. Blood glucose will be measured every five minutes for the first approximately 2.5 hours, and thereafter every 10-15 minutes. During the glucose-clamp study day the infusion rate of glucose will be adjusted continuously to match the glucose levels measured on the glucagon study day.

Blood samples for the analysis of plasma glucagon, insulin, C-peptide etc. will be drawn every five minutes for the first 60 minutes, and thereafter every 15-30 minutes.

After approximately three hours cognitive testing will be performed. After four hours, the infusion of either glucagon or glucose will be terminated. The final blood samples will be drawn 15 and 30 minutes after termination of the infusion.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the participant information and signing the consent form
* Between 25 and 70 years of age at the time of screening
* Body mass index (BMI) ≤ 25 kg/m2 at the time of screening
* A minimum of 7 years of schooling

Exclusion Criteria:

* Enrolment in other research projects that might interfere with the study
* Diabetes diagnosis (type 1 and 2)
* Pregnancy or breastfeeding
* Use of medications which, in the opinion of the investigator, may jeopardise participant's safety or compliance with the protocol
* Diagnosis of psychiatric disorders, dementias, or any other neurological disorders that in the opinion of the investigator precludes compliance with the study protocol, evaluation of the results or represents an unacceptable risk for the participants safety
* Severe claustrophobia
* Impaired liver function defined as either alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) ≥ 2 times normal values
* Kidney disease defined as serum creatinine levels ≥ 126 μmol/L for male and ≥ 111 μmol/L for female
* Cardiac problems including any of the following:

  1. Classified as being in New York Heart Association (NYHA) class III or IV
  2. Angina pectoris (chest pain) within the last 6 months
  3. Acute myocardial infarction (heart attack) within last 2 years
* Inadequately treated blood pressure at screening defined as repeated resting blood pressure outside the range 90-150 mmHg for systolic and 50-100 mmHg for diastolic
* Active or recent malignant disease
* Inability to perform neuropsychological tests judged by the investigator (e.g. visual or auditory impairment or language barriers)
* Current or history of severe alcohol use or drug/chemical abuse as per investigator's judgement
* Any chronic disorders or severe diseases which, in the opinion of the investigator, might jeopardise participant's safety or compliance with the protocol

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
C-peptide (0-90 minutes) | During intervention (0-90 minutes)
  Difference in plasma concentrations of C-peptide assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day

SECONDARY OUTCOMES:
C-peptide to glucose ratio (0-90 minutes) | During intervention (0-90 minutes)
  Difference in plasma concentration of C-peptide assessed as area under the curve divided by plasma concentration of glucose assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day
C-peptide to glucose ratio (0-240 minutes) | During intervention (0-240 minutes)
  Difference in plasma concentration of C-peptide assessed as area under the curve divided by plasma concentration of glucose assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day
C-peptide (0-240 minutes) | During intervention (0-240 minutes)
  Difference in plasma concentrations of C-peptide assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day
C-peptide (0 minutes-glucose peak) | During intervention (0-time to plasma glucose peak concentration (assessed up to two hours))
  Difference in plasma concentrations of C-peptide assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day
C-peptide deconvolution (0-240 minutes) | During intervention (0-240 minutes)
  Difference in deconvolution of plasma concentrations of C-peptide between the glucagon infusion study day and the glucose clamp study day
Insulin (0-90 minutes) | During intervention (0-90 minutes)
  Difference in plasma concentrations of insulin assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day
Insulin (0-240 minutes) | During intervention (0-240 minutes)
  Difference in plasma concentrations of insulin assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day
Time to glucagon peak | During intervention (0-240 minutes)
  Time to glucagon peak on the glucagon study day
Time to glucagon steady state | During intervention (0-240 minutes)
  Time to glucagon steady state on the glucagon study day
Glucagon concentration at steady state | During intervention (0-240 minutes)
  Plasma glucagon steady state concentration on the glucagon infusion study day
Glucose (0-90 minutes) | During intervention (0-90 minutes)
  Difference in plasma glucose assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day
Glucose (0-240 minutes) | During intervention (0-240 minutes)
  Difference in plasma glucose assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day
Glucose peak | During intervention (0-240 minutes)
  Difference in plasma glucose peak concentration between the glucagon infusion study day and the glucose clamp study day
Time to glucose peak | During intervention (0-time to plasma glucose peak concentration (assessed up to two hours)
  Difference in time to plasma glucose peak concentration between the glucagon infusion study day and the glucose clamp study day
Glucose infused | During intervention (0-240 minutes)
  Glucose (g) infused on the glucose clamp study day
cAMP (0-90 minutes) | During intervention (0-90 minutes)
  Difference in plasma concentration of cAMP assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day
cAMP (0-240 minutes) | During intervention (0-240 minutes)
  Difference in plasma concentration of cAMP assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day
cAMP (240-300 minutes) | During intervention (240-300 minutes)
  Difference in plasma concentration of cAMP assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day
Cognitive function | During intervention (180-240 minutes)
  Difference in cognitive function assessed as a composite score from the cognitive testing (SCIP testing) between the glucagon infusion study day and the glucose clamp study day

OTHER OUTCOMES:
Word recall cognitive test | During intervention (180-240 minutes)
  Difference in the word recall cognitive test between the glucagon infusion study day and the glucose clamp study day
Three-letter recall cognitive test | During intervention (180-240 minutes)
  Difference in the three-letter recall cognitive test between the glucagon infusion study day and the glucose clamp study day
Verbal fluency cognitive test | During intervention (180-240 minutes)
  Difference in the verbal fluency cognitive test between the glucagon infusion study day and the glucose clamp study day
Delayed word recall cognitive test | During intervention (180-240 minutes)
  Difference in the delayed word recall cognitive test between the glucagon infusion study day and the glucose clamp study day
Visuomotor cognitive test | During intervention (180-240 minutes)
  Difference in the visuomotor cognitive test between the glucagon infusion study day and the glucose clamp study day
Triglycerides (0-240 minutes) | During intervention (0-240 minutes)
  Difference in plasma concentration of triglycerides assessed as area under the curve between the glucagon infusion study day and the glucose clamp study day

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai J Wewer Albrecthsen, MD PhD, Principal Investigator — Department of Clinical Biochemistry, Copenhagen University Hospital - Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark
Locations (1):
- Department of Clinical Biochemistry, Copenhagen University Hospital - Bispebjerg and Frederiksberg, Copenhagen, Denmark, Copenhagen, Denmark